CLINICAL TRIAL: NCT04242875
Title: Evaluation of Angle Kappa and Different Intraocular Lens Calculation Formulas in Acrysof® IQ Panoptix Intraocular Lens Outcomes, Visual Disturbances and Patient Satisfaction
Brief Title: The Effects of Angle Kappa on Clinical Outcomes With the PanOptix Intraocular Lens
Status: Completed | Type: Observational
Sponsor: Carolina Eyecare Physicians, LLC (Other)
Collaborators: Science in Vision (Other)
Responsible Party: Sponsor
Other Study IDs: CEP19-001
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Results first posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2022-06

CONDITIONS: Pseudophakia
MeSH Terms: conditions — Pseudophakia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- PanOptix: Participants will receive the PanOptix intraocular lens.
  Interventions: Diagnostic Test: Angle Kappa; Other: Visual disturbance questionnaire.

INTERVENTIONS:
Diagnostic Test: Angle Kappa — Angle kappa will be measured using the OPD III scan.
Other: Visual disturbance questionnaire. — Questionnaire evaluating visual disturbances.

SUMMARY:
Angle Kappa is considered a potential factor in explaining suboptimal outcomes with intraocular lenses (IOLs), particularly multifocal IOLs. Some evidence suggests this is not the case. This study was designed to investigate correlations between angle kappa and post-surgical outcomes with a trifocal IOL.

DETAILED DESCRIPTION:
The main complaint of patients who received a presbyopia correcting lens (regardless of the design) are visual disturbances such as glare, halos (rings around lights), starbursts (rays around light sources), mainly at night. The degree of limitation or how bothered patients are varies from patient to patient. To explain these symptoms different theories have been proposed including splitting the light into different focal points which decreases the intensity of the light reaching the retina. Most factors are common to all patients who received the lens; however, patients are not equally affected by these symptoms. Angle kappa has been considered a factor. Angle κ is the angle between the visual axis (straight line that passes through both the center of the pupil and the center of the fovea) and the pupillary axis (perpendicular line to the surface of the cornea that passes through the center of the pupil).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is undergoing bilateral lens extraction with intraocular lens implantation (PanOptix lens).
2. Willing and able to provide written informed consent for participation in the study
3. Willing and able to comply with scheduled visits and other study procedures.
4. Scheduled to undergo standard cataract surgery with topical anesthesia in both eyes within 6 to 30 days between surgeries.
5. Subjects who require an IOL power in the range of +6.0 D to +30.0 D only.
6. Subjects who require a TFNT00 or TFNT30 to TFNT60 IOL.
7. Potential postoperative visual acuity of 0.2 logMAR (20/32 Snellen) or better in both eyes.

Exclusion Criteria:

1. Severe preoperative ocular pathology
2. Subjects who require a higher toric power than the one available (TFNT60).
3. Uncontrolled diabetes.
4. Use of any systemic or topical drug known to interfere with visual performance.
5. Contact lens use during the active treatment portion of the trial.
6. Any concurrent infectious/non-infectious conjunctivitis, keratitis or uveitis.
7. Clinically significant corneal dystrophy
8. History of chronic intraocular inflammation.
9. History of retinal detachment.
10. Pseudoexfoliation syndrome or any other condition that has the potential to weaken the zonules.
11. Previous ocular surgery.
12. Severe dry eye
13. Pupil abnormalities
14. Anesthesia other than topical anesthesia (i.e. retrobulbar, general, etc).
15. Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or may interfere with the interpretation of study results.
16. Participation in (or current participation) any ophthalmic investigational drug or ophthalmic device trial within the previous 30 days prior to the start date of this trial.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing bilateral lens extraction and implantation of the presbyopia correcting lens PanOptix.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Solomon, Principal Investigator — Carolina Eyecare Physicians
Locations (1):
- Carolina Eyecare Physicians, LLC, Mt. Pleasant, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | PanOptix
Started | 30; 60 Eyes
Completed | 28; 56 Eyes
Not Completed | 2; 4 Eyes
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Arm/Group | PanOptix
Number analyzed (Participants) | 30
Number analyzed (Eyes) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
Angle Kappa [Mean (Standard Deviation); unit: mm] | 0.29 (0.17)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Angle Kappa in Visual Disturbances
Description: Frequency of visual disturbances with magnitude of Angle Kappa
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Groups:
- AK < 0.3 mm: Angle Kappa magnitude < 0.3 mm
- AK > 0.3 and <= 0.4 mm: Angle kappa magnitude > 0.3mm and <= 0.4mm
- AK > 0.4 mm: Angle kappa magnitude > 0.4mm
Arm/Group | AK < 0.3 mm | AK > 0.3 and <= 0.4 mm | AK > 0.4 mm
Number analyzed (Participants) | 10 | 6 | 12
Participants
  Glare frequency: Never | 4 | 4 | 5
  Glare frequency: Rarely | 1 | 0 | 0
  Glare frequency: Sometimes | 3 | 2 | 5
  Glare frequency: Most of the time | 0 | 0 | 2
  Glare frequency: Always | 2 | 0 | 0
  Halos frequency: Never | 3 | 4 | 3
  Halos frequency: Rarely | 0 | 0 | 1
  Halos frequency: Sometimes | 3 | 2 | 5
  Halos frequency: Most of the time | 1 | 0 | 2
  Halos frequency: Always | 3 | 0 | 1
  Starburst frequency: Never | 1 | 3 | 6
  Starburst frequency: Rarely | 0 | 0 | 0
  Starburst frequency: Sometimes | 3 | 3 | 5
  Starburst frequency: Most of the time | 2 | 0 | 1
  Starburst frequency: Always | 4 | 0 | 0

2. Secondary Outcome: Satisfaction With Vision by Magnitude of Angle Kappa
Description: Overall satisfaction score after surgery, categorized by magnitude of angle kappa
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Groups:
- AK > 0.3 mm and <= 0.4 mm: Angle kappa magnitude > 0.3 mm and <= 0.4 mm
- AK > 0.4 mm: Angle kappa magnitude > 0.4 mm
Arm/Group | AK < 0.3 mm | AK > 0.3 mm and <= 0.4 mm | AK > 0.4 mm
Number analyzed (Participants) | 10 | 6 | 12
Participants
  Very dissatisfied | 0 | 1 | 0
  Dissatisfied | 0 | 0 | 0
  Neither satisfied nor dissatisfied | 1 | 0 | 1
  Satisfied | 3 | 1 | 2
  Very satisfied | 6 | 4 | 9

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | PanOptix
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT04242875/Prot_SAP_000.pdf